CLINICAL TRIAL: NCT02362984
Title: The Role of DLBS1033 in the Management of Acute Ischemic Stroke Patients: A Randomized Controlled Study
Brief Title: DLBS1033 for the Treatment of Acute Ischemic Stroke
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Major technical hindrance in recruitment.
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS1033-0614
Record Dates: First submitted 2015-02-03; First posted 2015-02-13 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Acute Ischemic Stroke
Keywords: DLBS1033; acute ischemic stroke; MRS; mNIHSS
MeSH Terms: conditions — Ischemic Stroke | interventions — DLBS 1033

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): Placebo will be administered orally, 3 x 1 tablet daily, for 8 days of study period
  Interventions: Drug: Placebo
- DLBS1033 Group (Experimental): DLBS1033 will be administered orally, 3 x 1 tablet daily, for 8 days of study period
  Interventions: Drug: DLBS1033

INTERVENTIONS:
Drug: Placebo — Placebo of DLBS1033 will be given in addition to the standard therapy consisting of: aspirin enteric-coated tablet 1 x 80 mg daily, simvastatin film-coated tablet 1 x 20 mg daily, vitamin B complex 1 x 1 tablet daily, and citicholine injection 250 mg/2 mL twice daily
  Other Names: Placebo of DLBS1033
  Arms: Control Group
Drug: DLBS1033 — DLBS1033 enteric-coated tablets will be given in addition to the standard therapy consisting of: aspirin enteric-coated tablet 1 x 80 mg daily, simvastatin film-coated tablet 1 x 20 mg daily, vitamin B complex 1 x 1 tablet daily, and citicholine injection 250 mg/2 mL twice daily
  Other Names: Disolf
  Arms: DLBS1033 Group

SUMMARY:
This is a prospective, randomized, double-blind, and controlled clinical study to investigate the effects of DLBS1033 in conjunction with standard therapy compared to standard therapy alone in acute ischemic stroke patients.

DETAILED DESCRIPTION:
Patients included into the study will be randomized into two groups and receive either standard therapy alone (as control group) or standard therapy plus DLBS1033 at a dose of 490 mg three times daily (as DLBS1033 group). Standard therapy used in the study will consist of: aspirin 80 mg, simvastatin 20 mg, vitamin B complex, and citicholine 250 mg/2 mL twice daily.

After hospital admission and diagnosis, patient will be handled according to the standard management for acute ischemic stroke applicable in the hospital. Right after the patient is confirmed eligible to the study, the treatment(s) will be switched immediately into the study's regimens. Clinical and laboratory examinations to evaluate the investigational drug's efficacy will be performed at baseline, day 4, and day 8 of treatment (end of study); while safety examinations will be performed at baseline and end of study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with age of 18-75 years .
* Has been diagnosed with acute ischemic stroke clinically confirmed by CT scan.
* Modified National Institutes of Health Stroke Scale (mNIHSS) score >= 5.
* Patients present at hospital and receiving first dose of study medication within 72 hours after the onset of the stroke symptoms.
* Able to take oral medication.

Exclusion Criteria:

* For females of childbearing potential: pregnancy and lactation period.
* History of or current hemorrhagic stroke (within the last 3 months).
* Transient ischemic stroke (TIA).
* Patients with seizure at the onset of stroke.
* History of serious head injury within the last 3 months.
* History of major surgery within the last 3 months.
* Serious cardiovascular conditions, such as myocardial infarction, CHF grade III and IV (NYHA classification), aorta dissection, and atrial fibrillation within the last 6 months.
* Presence of severe renal or hepatic dysfunction
* Presence of acute or chronic infections.
* Thrombocytopenia (thrombocytes level < 150.000/ul).
* Patients with higher risks of bleeding.
* Uncontrolled hypertension (systolic blood pressure > 185 mmHg or diastolic blood pressure > 110 mmHg).
* Random plasma glucose >= 200 mg/dL.
* Current or regular use of oral anticoagulants, antiplatelets other than study medication, and herbal medicines.
* Hypersensitive to the investigational product(s).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Improvement in mNIHSS score | 7 days after treatment initiation
  Change in functional outcomes as measured by The Modified National Institute of Health Stroke Scale (mNIHSS) from its baseline value

SECONDARY OUTCOMES:
Improvement in MRS | 7 days after treatment initiation
  Change in functional outcomes as measured by Modified Rankin Scale (MRS) from its baseline value
Improvement in fibrinogen level | 7 days after treatment initiation
  Change in haemostatic parameter as measured by fibrinogen level from its baseline value
Improvement in d-dimer level | 7 days after treatment initiation
  Change in haemostatic parameter as measured by d-dimer level from its baseline value
Liver function | 7 days after treatment initiation
  Liver function measured will be: serum AST, ALT, G-GT, total bilirubin
Renal function | 7 days after treatment initiation
  Renal function measured will be serum creatinine
Routine hematology | 7 days after treatment initiation
  Routine hematology measured will be: hemoglobin, hematocrit, RBC, WBC, differentiation of WBC, and platelet count
Hemostasis parameters | 7 days after treatment initiation
  Hemostasis parameters measured will be: PT and aPTT
Adverse events | 7 days after treatment initiation
  Adverse events, including bleeding events, will be observed and carefully evaluated during the expected average of 7 days of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tut W Handayani, Sp.S, MD, Principal Investigator — RSUD R. Syamsudin, SH
Locations (1):
- RSUD R. Syamsudin, SH, Sukabumi, West Java, Indonesia